CLINICAL TRIAL: NCT02374151
Title: Accuracy of Electrohysterography in Assessing Intrauterine Pressure Compared to Invasive Intrauterine Pressure Catheter
Brief Title: Accuracy of Electrohysterography in Assessing Intrauterine Pressure
Acronym: EHG
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Aya Mohr Sasson, Sheba Medical Center
Other Study IDs: 1980- 15-SMC
Record Dates: First submitted 2015-02-22; First posted 2015-02-27 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Uterine Pressure Measurement
Keywords: intrauterine pressure catheter; electrohysterography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with IUPC: Women at term in second or third phase of labor who are indicated to have an IUPC during active labor
  Interventions: Device: Electrohysterography

INTERVENTIONS:
Device: Electrohysterography — The EHG uses a Graphium electrode patch that is applied to the abdomen and records electrical activity non-invasively
  Other Names: PureTrace

SUMMARY:
This is a case control prospective study aiming to investigate the accuracy of the electrohysterography (EHG) compared to the intrauterine pressure catheter ( IUPC) that is commonly used in delivery room. Women in second phase of labor - indicated for insertion of IUPC will be asked to participate . Patients that will give their informed consent will be connected both to IUPC and EHG. Medical history and demographic parameters will be taken. The graphs will be compared and analyzed for its frequency and intensity. Delivery mode and fetal well-being will be recorded

DETAILED DESCRIPTION:
Fetal monitoring relies on sensors to measure uterine activity and fetal heart rate. Monitoring contractions during labor using the external tocodynamometer relies on measurement of the activity of the abdominal wall and is sometimes unreliable and inaccurate .In cases that there is difficulty in monitoring uterine wall activity through the abdominal wall or increased risk for uterine wall rupture, the commonly used alternative is an invasive intrauterine pressure catheter monitor (IUPC). The IUPC is applied gently behind the head of the fetus after rupture of the membranes spontaneously or artificially into the uterine cavity. Insertion of IUPC monitor may be associated with rare but serious complications including placental abruption and uterine rupture. Non invasive method that will allow for accurate and precise monitoring of the uterine muscle activity is well under search

Lately, a new electrohysterography (EHG) device was introduced as an alternative to the standard intrauterine sensors. (Nemo Healthcare's, Netherlands, PUREtrace). When muscle cells contract, small changes occur in the electrical potential across the cell walls. During contractions, the electrical activity of the uterine muscle can be measured on the maternal abdomen. EHG has been developed to measure the electrical muscle activity of the uterus directly, and by that claiming to offer highly accurate information that correlates with existing invasive measurement methods for uterine contractions. Vlemminx et al, showed EHG also appears to report a more detailed tocographic waveform, like hypertonia or unorganized electrical uterine activity.

The EHG uses a Graphium electrode patch that is applied to the abdomen and records electrical activity non-invasively. Its' module amplifies and converts these signals to a recognized measurement method for uterine activity, as commonly used in fetal monitoring. This measurement is independent of the Body-Mass-Index, abdominal wall thickness or maternal position enabling monitoring obese patients as well.

By using the Graphium electrode patch the patient comfort increases significantly when compared to other measurement methods. The patch is also easy to apply for the medical staff and does not require repositioning over time. It provides a safe and patient-friendly alternative for measuring uterine activity, without the need of changing the existing fetal monitoring infrastructure.

The aim of this study is to investigate the accuracy of the electrohysterography compared to the intrauterine pressure catheter that is commonly used in delivery room in order to promote less invasive management protocols in the future in order to better predict uterine muscle dysfunction during labor.

This is a case control prospective study. Women in second phase of labor - indicated for insertion of intrauterine pressure catheter due to previous uterine scar, multifetal pregnancy, grand multiparity or dysfunctional labor will be asked to participate . Patients that will give their informed consent to participate in the study, will be connected both to IUPC and EHG.Medical history and demographic parameters will be taken. The graphs will be compared and analyzed for its frequency and intensity. Delivery mode and fetal well-being will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Women at term in second or third phase of labor who are indicated to have an IUPC during active labor

Exclusion Criteria:

* Women not in labor
* Active skin disease

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women at term in second or third phase of labor who are indicated to have an IUPC during active labor
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of uterine contraction sensing, comparing to invasive intrauterine catheter. | From insertion of IUPC untill its' removal ( due to vaginal delivery or referral to instrumental/ caesarean delivery).

SECONDARY OUTCOMES:
Final delivery mode | Third phase of delivery
  spontaneous, instrumental, caesarean

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr Sasson, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- See also: article describing the benefit of the electrohysterography — http://www.medscape.com/medline/abstract/25650036
- See also: The company internet site — http://www.nemohealthcare.com/en/